CLINICAL TRIAL: NCT03772184
Title: Alalfy Modofied Cervical Inversion During CS in Placenta Previa
Brief Title: Modified Cervical Inversion During CS in Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Collaborators: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Lecturer Obstetrics and Gyneology , National Research Centre, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Modified cervical inversion
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Intervention Model Description: Using cervical inversion during cesarean section
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical inversion (Active Comparator)
  Interventions: Procedure: Cervical inversion
- no cervical inversion (No Intervention)

INTERVENTIONS:
Procedure: Cervical inversion — inverting the cervical lip after delivery
  Arms: cervical inversion

SUMMARY:
There is an increasing rates of placenta previa nowadays

DETAILED DESCRIPTION:
several techniques were described to control bleeding .

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 38 weeks or more with placenta previa

Exclusion Criteria:

* pregnant ladies with normally implanted placenta or placenta accreat , increta or percreta

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women with placenta previa
Enrollment: 240 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
The number of women whose placental bed bleeding will be controlled by cervical inversion cervical inversion | within an hour
  how can the cervical inversion technique controls the placental bed bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — National research centre , Aljazeerah hospital
Locations (1):
- Algazeerah and helwan university, Giza, Egypt